CLINICAL TRIAL: NCT04693286
Title: A Phase II Clinical Trial to Evaluate the Safety and Immunogenicity of Novel Oral Polio Type 2 Vaccine Candidate in Healthy Newborns in Bangladesh
Brief Title: Clinical Trial of Novel OPV2 Vaccine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); Centers for Disease Control and Prevention (U.S. Federal Agency); PATH (Other); World Health Organization (Other); PT Bio Farma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PR-20001
Record Dates: First submitted 2020-12-14; First posted 2021-01-05 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-02

CONDITIONS: Poliomyelitis
Keywords: Safety; Immunogenecity; nOPV2; Newborn; Bangladesh
MeSH Terms: conditions — Poliomyelitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vaccine candidate arm (Active Comparator): In this arm, participants will get nOPV2 vaccine candidate 1
  Interventions: Biological: novel oral polio type 2 vaccine (nOPV2)
- Placebo arm (Placebo Comparator): In this arm, participants will get inactive substance like sucrose in BME media and buffer.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: novel oral polio type 2 vaccine (nOPV2) — • nOPV2 (C1) is a live-attenuated serotype-2 poliovirus that was derived from a modified Sabin type-2 infectious cDNA clone and propagated in Vero cells (S2/cre5/S15domV/rec1/hifi3). Placebo contain sucrose in buffer.
  Arms: Vaccine candidate arm
Other: Placebo — Placebo contains no active ingradients, only sucrose in buffer
  Arms: Placebo arm

SUMMARY:
Though OPV is safe and effective, it can mutate and reacquire neurovirulence in rare circumstances. This can result in vaccine-associated paralytic polio and circulating vaccine-derived polioviruses. Use of tOPV had risk of generating VAPP and seeding new type 2 circulating vaccine-derived polioviruses though wild type 2 virus was eradicated in September 2015. For this reason tOPV vaccine was withdrawn globally in April 2016 and switched to bOPV. cVDPV2 outbreaks have occurred in sixteen countries after cassation of OPV2. Using stockpiled mOPV2 to respond to this situation risks propagating new cVDPVs. IPV induces only limited intestinal mucosal immunity not effective to interrupt fecal-oral route transmission in settings of poor hygiene and sanitation. Therefore, development of novel oral polio vaccine with enhanced genetic stability and lower risk of reversion to neurovirulence compared to current Sabin 2 strains is major priority of global polio eradication Program

Current clinical development plan outlines studies through Phase II development with nOPV2 candidate strains being tested in adult toddler and infant populations who received prior dose of OPV or IPV. No study has been conducted in truly naive newborns with no prior receipt of any polio vaccines

Hypothesis: Vaccinating healthy newborns with novel type 2 polio virus candidate vaccines is safe and can induce putatively protective immune response

Objectives

Primary Objective

Safety

To evaluate the safety and tolerability after one and two doses of nOPV2 vaccine candidates 1 given 4 weeks apart in poliovirus vaccine-naïve newborn Immunogenicity To evaluate the immune response to vaccination after one and two doses of nOPV2 vaccine candidate 1 given 4 weeks apart in poliovirus vaccine-naïve newborns

Secondary objectives

Immunogenicity

To evaluate seroprotection rate geometric mean and median titers to vaccination after one dose of nOPV2 vaccine candidate 1 in poliovirus vaccine-naïve newborns To further evaluate seroprotection rate geometric mean and median titers to vaccination after two doses of nOPV2 candidate 1 in poliovirus vaccine-naïve newborns

Viral Shedding

To assess trate of fecal viral shedding at fixed time points following one and two doses of nOPV2 vaccine candidate 1 in newborns To assess duration of fecal viral shedding at fixed time points following one and two doses of nOPV2 vaccine candidate 1 in newborns To assess extent of fecal viral at fixed time points following one and two doses of nOPV2 vaccine candidate 1 in newborns

Exploratory objective

To assess genetic stability through genetic deep sequencing assay and neurovirulence test through transgenic mice NV assays from a subset of participants stools samples

DETAILED DESCRIPTION:
Burden: Oral Polio Vaccine (OPV) contains attenuated (weakened) polioviruses. Though OPV is safe and effective, it can mutate and reacquire neurovirulence in rare circumstances. This can result in vaccine-associated paralytic polio (VAPP) and circulating vaccine-derived polioviruses (cVDPVs) on rare occasions. Use of tOPV, therefore, had the risk of generating VAPP and seeding new type 2 circulating vaccine-derived polioviruses (cVDPV2), even though the wild type 2 virus was eradicated in September 2015. For this reason tOPV vaccine was withdrawn globally in April 2016 and switched to the bivalent oral poliovirus vaccine (bOPV). Circulating vaccine-derived type-2 poliovirus (cVDPV2) outbreaks have occurred in sixteen countries after cassation of OPV2. Using stockpiled mOPV2 to respond to this situation risks propagating new cVDPVs and this phenomenon has already been observed in multiple geographies following the switch. Inactivated polio vaccine (IPV) induces only limited intestinal mucosal immunity and is not effective to interrupt fecal-oral route transmission in settings of poor hygiene and sanitation. Therefore, development of novel oral polio vaccine/s with enhanced genetic stability and lower risk of reversion to neurovirulence compared to current Sabin 2 strains is a major priority of the global polio eradication Program.

Knowledge gap: The current clinical development plan outlines studies through Phase II development with the nOPV2 candidate strains being tested in adult, toddler, and infant populations who have received prior dose/s of OPV and/or IPV. No study has been conducted in truly naive newborns with no prior receipt of any polio vaccines to strengthen the clinical evidence in favour of utilizing these novel OPV strains.

Relevance: Existing Sabin type 2 polio virus vaccines can mutate in to pathogenic virus and become neurovirulent, causing VAPP and cVDVP. So novel type 2 polio virus candidate vaccines is an urgent need especially for outbreak situations. The nOPV2 strains are intended for use as safer alternatives to mOPV2 vaccines for outbreak response. Data from this proposed study result will further strengthen the clinical evidence base to deploy novel, genetically stable OPV strains to reduce the risk of generating cVDPV and VAPP. The study will generate data on novel OPV2 candidates for pre-licensure use in outbreak scenarios and for eventual full licensure and WHO Prequalification.

Hypothesis : Vaccinating healthy newborns with novel type 2 polio virus candidate vaccines (nOPV2) is safe and can induce a putatively protective immune response.

Objectives:

Primary Objectives:

Safety:

• To evaluate the safety and tolerability after one and two doses of nOPV2 vaccine candidates 1, given 4 weeks apart in poliovirus vaccine-naïve newborns.

Immunogenicity:

• To evaluate the immune response (measured by seroconversion rate) to vaccination after one and two doses of nOPV2 vaccine candidate 1, given 4 weeks apart in poliovirus vaccine-naïve newborns.

Secondary objectives:

Immunogenicity:

* To evaluate seroprotection rate, geometric mean and median titers to vaccination after one dose of nOPV2 vaccine candidate 1 in poliovirus vaccine-naïve newborns.
* To further evaluate seroprotection rate, geometric mean and median titers to vaccination after two doses of nOPV2 candidate 1 in poliovirus vaccine-naïve newborns.

Viral Shedding:

* To assess the rate of fecal viral shedding (as determined by real-time RT-PCR) at fixed time points following one and two doses of nOPV2 vaccine candidate 1 in newborns.
* To assess the duration of fecal viral shedding (as determined by real-time RT-PCR) at fixed time points following one and two doses of nOPV2 vaccine candidate 1 in newborns.
* To assess the extent of fecal viral shedding ( the quantity of nOPV2 virus shedding, measured asCCID50 per g of stool) at fixed time points following one and two doses of nOPV2 vaccine candidate 1 in newborns.

Exploratory objective:

• To assess genetic stability through genetic deep sequencing assay and neurovirulence test through transgenic mice NV assays from a subset of participants stools samples.

Methods:

The study is a Phase II clinical trial which will be conducted in rural Bangladesh at Matlab. The total enrolment target for the clinical trial is 330 , with 220 in nOPV2 candidate 1 arm and 110 in placebo arm. All participants will be randomized (in block randomization of variable length) 2:1 ratio to nOPV2 vaccine candidate C1(2 drops) and placebo group (2 drops). All eligible healthy newborn participants will be vaccinated orally at birth and at 4 weeks of age with C1 (105.0± 0.5 CCID50, 2 drops) or placebo (2 drops) of age followed by fIPV + bOPV at week 8, bOPV at week 12 and fIPV + bOPV at week 16 and other vaccines according to EPI schedule in Bangladesh.

In order to record any immediate reaction participants will be observed for 30 minutes following each dose of vaccination. Study staff will visit homes of the participants daily for 7 days to collect systemic solicited adverse events after study vaccination using electronic dairy cards. Unsolicited adverse events, adverse events of special interest and serious adverse events will be collected throughout the entire study period by weekly home visit. Mothers of the participant will be provided a telephone number to communicate with the investigator for any adverse or serious adverse events.

Three blood samples each of 1 ml, will be collected to measure the immune response of nOPV vaccine candidate 1: the first pre-vaccine blood sample on the day of first dose nOPV2 vaccine candidate 1 /placebo (at birth), second blood sample at 4 weeks before second dose nOPV2 vaccine candidate 1 /placebo and the third blood sample will be collected at 8 weeks before giving fIPV + bOPV vaccine.

Mothers of enrolled participants will be requested to collect about 8 grams (about the size of one adult thumb) of stool from participants to assess viral sheddings. A total of seven stool samples will be collected: the first pre-vaccine sample will be collected on the day of first dose nOPV2 vaccine candidate 1 /placebo (at birth), second sample at week 2, third sample at week 4 before second dose nOPV2 vaccine candidate 1 /placebo, fourth stool sample at week 6, fifth stool at week 8 before giving fIPV + bOPV vaccine, sixth stool sample at week 10 and seventh sample at week 12 of age to assess viral shedding.

Outcome measures/variables:

Safety

* Incidence rate of solicited systemic AEs within 7 days after each dose of vaccine
* Incidence rate of unsolicited AEs during entire study period
* Incidence rate of serious AEs and AESIs during entire study period

Immunogenicity

* Seroconversion rate as measured by microneutralization assay (MN) for OPV Type 2
* Seroprotection rate as measured as seropositivity by MN for OPV Type 2
* Geometric mean and median titers as measured by MN for OPV Type 2

Viral Shedding

* Rate of fecal viral shedding by real-time RT-PCR
* Duration of fecal viral shedding by real-time RT-PCR
* Extent of fecal viral shedding ( the quantity of nOPV2 virus shedding, measured as CCID50 per g of stool) at fixed time points following different dose schedule.

Genetic stability

• Genetic deep sequencing assay and neurovirulence test through transgenic mice NV assays from a subset of participants stools samples.

ELIGIBILITY:
Inclusion Criteria:

* Newborns at birth (range: 0-3 days of age).
* Mothers that consent for participation in the full length of the study.
* Mothers those are able to understand and comply with planned study procedures.

Exclusion Criteria:

* Mother and newborns who are unable to participate in the full length of the study.
* A diagnosis or suspicion of immunodeficiency disorder either in the newborn or in an immediate family member.
* A diagnosis or suspicion of bleeding disorder that would contraindicate collection of blood by venipuncture.
* Acute diarrhea, infection or illness at the time of enrollment that would require admission to a hospital.
* Acute vomiting and intolerance to liquids within 24 hours before the enrollment visit.
* Receipt of any polio vaccine (OPV or IPV) and Rotavirus Vaccine (RVV) before enrollment based upon documentation or mothers recall.
* Newborns from multiple births. Newborns from multiple births will be excluded to reduce the potential for contact transmission of vaccine poliovirus to siblings. The newborn from a multiple birth who is /are not enrolled would be likely to receive routine immunization and transmit vaccine poliovirus to the enrolled infant.
* Newborns from premature births (<37 weeks of gestation).

Ages: 1 Hour to 3 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 330 (Actual)
Dates: Start 2020-09-21 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Safety of nOPV2 vaccine | Upto 3 months
  * Incidence rate of solicited systemic AEs within 7 days after each dose of vaccine
  * Incidence rate of unsolicited AEs during entire study period
  * Incidence rate of serious AEs and AESIs during entire study period
Immunogenecity of nOPV2 vaccine , will be assessed as poliovirus type-2-specific serum neutralising antibodies | 4 weeks
  Proportion of participants showing seroconversion and seroprotection will be calculated and reported
Viral shedding in participants stool will be measured and reported by proportion of participants showing viral shedding in their stools, the time to cessation of viral shedding, the cell culture infective dose of shed virus in virus-positive stools | 12 weeks
  Vaccine poliovirus shedding in the study participants stool will be assessed by real-time RT-PCR method.

SECONDARY OUTCOMES:
Genetic assay and Neurovirulance test to assess genetic stability by demonstrating the retention of key genetic regions engineered in the vaccine candidate | 4 weeks
  WHO poliovirus receptor transgenic mouse (Tg-PVR21) neurovirulence test will be used. Deep sequencing will be performed on the cell culture-amplified virus and on viral RNA isolated from participants

CONTACTS AND LOCATIONS:
Overall Officials: K Zaman, PhD FRCP, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (1):
- : International Centre for Diarrhoeal Disease Research, Bangladesh, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared with BMGF, PATH, CDC, WHO
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: July 2021

REFERENCES:
- [Derived] Godin A, Brickley EB, Connor RI, Wieland-Alter WF, Weiner JA, Ackerman ME, Modlin JF, Sajjad OM, Arita M, Gast C, Mainou BA, Zaman K, Hoque M, Rana S, Bandyopadhyay AS, Wright PF. Intestinal mucosal immune responses to novel oral poliovirus vaccine type 2 in healthy newborns. Clin Infect Dis. 2025 Sep 5:ciaf484. doi: 10.1093/cid/ciaf484. Online ahead of print. PMID 40907970
- [Derived] Zaman K, Bandyopadhyay AS, Hoque M, Gast C, Yunus M, Jamil KM, Mainou BA, Konopka-Anstadt JL, Hendley WS, Vincent A, Clemens R, Clemens SAC, Ross AG, Clemens JD, Tritama E. Evaluation of the safety, immunogenicity, and faecal shedding of novel oral polio vaccine type 2 in healthy newborn infants in Bangladesh: a randomised, controlled, phase 2 clinical trial. Lancet. 2023 Jan 14;401(10371):131-139. doi: 10.1016/S0140-6736(22)02397-2. Epub 2022 Dec 7. PMID 36495882